CLINICAL TRIAL: NCT01841983
Title: Project A: Integrated Approaches to Improving the Health and Safety of Health Care Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Partners HealthCare (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Boston University (Other); Carelon Research (Other)
Responsible Party: Principal Investigator, Glorian Sorensen, Professor of Society, Human Development, and Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: U19OH008861 (NIH)
Record Dates: First submitted 2013-03-19; First posted 2013-04-29 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Health Behavior; Sleep; MSDs; Dietary Habits; Physical Activity
Keywords: Total worker health; Sleep; MSDs; Diet; Physical Activity
MeSH Terms: conditions — Health Behavior; Feeding Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Be Well Work Well
  Interventions: Other: Be Well Work Well
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Be Well Work Well — The intervention follows principles for integrated approaches to promoting and protecting worker health. It will occur on 4 inpatient units at Massachusetts General Hospital beginning in January 2013, and will continue for 1 year.
  Overall intervention objectives:
  1. Motivate individual staff members to engage in targeted health and safety behavior changes;
  2. build awareness of ergonomic and safety hazards and of opportunities for healthy dietary choices and physical activity;
  3. facilitate unit-level norms supportive of breaks, safe patient handling, and targeted health and safety behaviors; and
  4. promote co-worker and supervisor support for targeted health and safety behaviors.
  Other Names: OSH protection and health promotion program
  Arms: Intervention

SUMMARY:
While most of the research on integrated approaches of occupational health and safety and worksite health promotion to date has focused on manufacturing settings, employment is shifting to the service sector. Within this sector, health care employs over 12 million workers, and is the second fastest growing industry in the U.S. economy. In contrast to workers in other industries, rates of occupational injuries and illnesses among health care workers have increased over the past decade. The purpose of this study is to lay the foundation for integrated interventions in health care through examination of the associations of worker health outcomes and risks on and off the job with work policies and practices and to address the prevalent issues of musculoskeletal disorders (MSDs), particularly low back pain disability (LBPD), and health promotions through physical activity among patient care workers. The specific aims of this study are:

1. To estimate the efficacy and determine the feasibility of an integrated intervention, addressing both health protection and health promotion in order to reduce MSD symptoms and improve health behaviors among healthcare workers. We will assess between-group differences in MSD symptoms, health behaviors, including physical activity, and a set of secondary outcomes, including unplanned absence, reported injuries, worker compensation claims and costs, turnover and retention, intention to leave the job, and work-role function. This study will explore the working hypothesis that: Workers employed at baseline in patient-care units receiving the intervention will report greater reductions in their MSD symptoms (primary outcome) and greater improvements in health behaviors, compared with workers employed at baseline in units assigned to the Usual Care control group.
2. To determine the factors in the work environment which contribute over time to reductions in MSD symptoms and improvements in safe and healthy behaviors. (1) The work environment, work organization, and psychosocial factors, measured in our current study, will be associated with changes in workers' health behaviors and health outcomes between the assessments in the current and proposed studies; (2) Improvements in the work environment over time will be associated with improvements in workers' health behaviors and health outcomes. We will conduct multilevel modeling analysis to evaluate the simultaneous effects of worker-level and unit-level factors on MSD symptoms and safety and health behaviors.

DETAILED DESCRIPTION:
Improving and protecting the health and well-being of healthcare workers requires addressing key risks in the work environment as well as promoting safe and healthy behaviors. Healthcare workers are at elevated risk for musculoskeletal disorders (MSDs) due to a range of job factors, including lifting and transferring patients; working long hours (often at night); and limited control over decisions on the job. Among these, nurses and nurses aides bear the largest burden of injury. Back injuries in particular constitute the greatest source of their disability. These risks are likely to increase in coming years due to the aging nursing workforce, increase in work demands, and labor shortages. Health behaviors, including physical activity, inadequate sleep, and dietary patterns associated with being overweight or obese, are also influenced by the work environment and psychosocial factors on the job, and are also associated with MSD risk. Traditional approaches to redressing these risks have focused separately on health protection, including efforts to reduce MSD risk, and health promotion aimed at improving health behaviors. Little research has systematically examined the dual and potentially synergistic effects of the work environment on risk of MSDs and worker health behaviors, and there is insufficient evidence to determine the most efficacious ways to ameliorate the combined effects of these health risks. Our long-term goal is to improve the overall health and well-being of healthcare workers by making available evidence-based worksite policies, programs, and practices that foster a healthy work environment, reduce potential hazardous job exposures, and promote safe and healthy behaviors. The proposed study is the next logical step in building this evidence base. Factors in the work environment, including high work demands, low social support, and long work hours, have been shown to increase risk of MSDs, as well as risk-related behaviors. Yet little research has systematically explored these cross-cutting pathways and their implications for improving the effectiveness of worksite interventions to address the broad spectrum of worker health outcomes.

The proposed research provides a novel approach to worksite interventions that integrate occupational safety and health and worksite health promotion, taking into account the shared factors in the work environment shaping both MSDs and health behaviors. Standard approaches to occupational health and safety and worksite health promotion are based on a parallel structure of separate silos functioning relatively independently in the worksite, each drawing from their own disciplines and training experiences within public health. Although these parallel efforts share the common mission of improving worker health, their strategies are based on different assumptions about and approaches to improving worker health outcomes. The proposed research integrates these parallel approaches. Although our prior research has rigorously tested the efficacy of this integrated intervention model in changing worker health behaviors, to our knowledge no prior research has examined the impact of this integrated model on health outcomes associated with work exposures - here, notably, on MSD symptoms.

ELIGIBILITY:
Inclusion criteria:

* Adult and pediatric in-patient care units at Massachusetts General Hospital that have ceiling lifts in place (n=42 units) are eligible for the intervention.
* Patient care workers, including registered nurses (RNs), licensed practical nurses (LPNs), patient care assistants (PCAs)/nursing assistants (NAs) and Nurse Leaders working in in-patient units for at least 20 hours per week (n= 9500).
* Of those patient care workers, those working in adult and pediatric in-patient care units (n=90 units) are eligible to be randomly selected for surveys.

Exclusion criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9500 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pain | Baseline and 1 year
  * Musculoskeletal disorder pain
  * Self-report via survey
Physical Activity | Baseline and 1 year
  Self-report via survey
Diet | Baseline and 1 year
  Self-report via survey
Sleep | Baseline and 1 year
  Self-report via survey

SECONDARY OUTCOMES:
Safe patient handling | Baseline and 1 year
  Self-report via survey
Work role function/limitations | Baseline and 1 year
  Self-report via survey
BMI/obesity | Baseline and 1 year
  Self-report via survey

OTHER OUTCOMES:
Economic/systems outcomes | Baseline and 1 year
  * Unplanned absence
  * Reported injuries
  * Worker compensation
  * Turnover/retention
  * Healthcare utilization/costs
  Self-report via survey

CONTACTS AND LOCATIONS:
Overall Officials: Glorian Sorensen, PhD, MPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Harvard School of Public Health, Boston, Massachusetts

REFERENCES:
- [Background] Sembajwe G, Tveito TH, Hopcia K, Kenwood C, O'Day ET, Stoddard AM, Dennerlein JT, Hashimoto D, Sorensen G. Psychosocial stress and multi-site musculoskeletal pain: a cross-sectional survey of patient care workers. Workplace Health Saf. 2013 Mar;61(3):117-25. doi: 10.1177/216507991306100304. PMID 23452130
- [Background] Kim SS, Okechukwu CA, Dennerlein JT, Boden LI, Hopcia K, Hashimoto DM, Sorensen G. Association between perceived inadequate staffing and musculoskeletal pain among hospital patient care workers. Int Arch Occup Environ Health. 2014 Apr;87(3):323-30. doi: 10.1007/s00420-013-0864-y. Epub 2013 Mar 12. PMID 23475312
- [Background] Sabbath EL, Hurtado DA, Okechukwu CA, Tamers SL, Nelson C, Kim SS, Wagner G, Sorenson G. Occupational injury among hospital patient-care workers: what is the association with workplace verbal abuse? Am J Ind Med. 2014 Feb;57(2):222-32. doi: 10.1002/ajim.22271. Epub 2013 Oct 22. PMID 24151093
- [Background] Caspi CE, Dennerlein JT, Kenwood C, Stoddard AM, Hopcia K, Hashimoto D, Sorensen G. Results of a pilot intervention to improve health and safety for health care workers. J Occup Environ Med. 2013 Dec;55(12):1449-55. doi: 10.1097/JOM.0b013e3182a7e65a. PMID 24270297
- [Background] Sorensen G, McLellan D, Dennerlein JT, Pronk NP, Allen JD, Boden LI, Okechukwu CA, Hashimoto D, Stoddard A, Wagner GR. Integration of health protection and health promotion: rationale, indicators, and metrics. J Occup Environ Med. 2013 Dec;55(12 Suppl):S12-8. doi: 10.1097/JOM.0000000000000032. PMID 24284762
- [Background] Umukoro PE, Arias OE, Stoffel SD, Hopcia K, Sorensen G, Dennerlein JT. Physical activity at work contributes little to patient care workers' weekly totals. J Occup Environ Med. 2013 Dec;55(12 Suppl):S63-8. doi: 10.1097/JOM.0000000000000046. PMID 24284756
- [Background] Nelson CC, Wagner GR, Caban-Martinez AJ, Buxton OM, Kenwood CT, Sabbath EL, Hashimoto DM, Hopcia K, Allen J, Sorensen G. Physical activity and body mass index: the contribution of age and workplace characteristics. Am J Prev Med. 2014 Mar;46(3 Suppl 1):S42-51. doi: 10.1016/j.amepre.2013.10.035. PMID 24512930
- [Result] Kim SS, Okechukwu CA, Buxton OM, Dennerlein JT, Boden LI, Hashimoto DM, Sorensen G. Association between work-family conflict and musculoskeletal pain among hospital patient care workers. Am J Ind Med. 2013 Apr;56(4):488-95. doi: 10.1002/ajim.22120. Epub 2012 Sep 27. PMID 23019044
- [Result] Hopcia K, Dennerlein JT, Hashimoto D, Orechia T, Sorensen G. Occupational injuries for consecutive and cumulative shifts among hospital registered nurses and patient care associates: a case-control study. Workplace Health Saf. 2012 Oct;60(10):437-44. doi: 10.1177/216507991206001005. Epub 2012 Sep 24. PMID 22998692
- [Result] Buxton OM, Hopcia K, Sembajwe G, Porter JH, Dennerlein JT, Kenwood C, Stoddard AM, Hashimoto D, Sorensen G. Relationship of sleep deficiency to perceived pain and functional limitations in hospital patient care workers. J Occup Environ Med. 2012 Jul;54(7):851-8. doi: 10.1097/JOM.0b013e31824e6913. PMID 22796931
- [Result] Reme SE, Dennerlein JT, Hashimoto D, Sorensen G. Musculoskeletal pain and psychological distress in hospital patient care workers. J Occup Rehabil. 2012 Dec;22(4):503-10. doi: 10.1007/s10926-012-9361-5. PMID 22466375
- [Result] Dennerlein JT, Hopcia K, Sembajwe G, Kenwood C, Stoddard AM, Tveito TH, Hashimoto DM, Sorensen G. Ergonomic practices within patient care units are associated with musculoskeletal pain and limitations. Am J Ind Med. 2012 Feb;55(2):107-16. doi: 10.1002/ajim.21036. Epub 2011 Nov 23. PMID 22113975
- [Result] Boden LI, Sembajwe G, Tveito TH, Hashimoto D, Hopcia K, Kenwood C, Stoddard AM, Sorensen G. Occupational injuries among nurses and aides in a hospital setting. Am J Ind Med. 2012 Feb;55(2):117-26. doi: 10.1002/ajim.21018. Epub 2011 Oct 24. PMID 22025077
- [Result] Sorensen G, Stoddard AM, Stoffel S, Buxton O, Sembajwe G, Hashimoto D, Dennerlein JT, Hopcia K. The role of the work context in multiple wellness outcomes for hospital patient care workers. J Occup Environ Med. 2011 Aug;53(8):899-910. doi: 10.1097/JOM.0b013e318226a74a. PMID 21775897
- See also: Center for Work, Health, and Wellbeing — http://centerforworkhealth.sph.harvard.edu/